CLINICAL TRIAL: NCT06497582
Title: Self-acupressure and Zhan Zhuang for Pain, Fatigue, and Sleep Disturbance in Breast Cancer Survivors: A Pilot Randomized Controlled Trial
Brief Title: Self-acupressure and Zhan Zhuang for Symptom Cluster Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 04
Record Dates: First submitted 2024-05-28; First posted 2024-07-12 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer Female; Survivorship

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Zhan-zhuang group (Experimental): The intervention will last 8 weeks and comprise the following
  1) Two sessions of Zhan Zhuang training(2 hours per session/week, totally 4 hours) for 2 weeks. (2) self-practice of zhan-zhuang for 6 weeks (daily, at least 20 mins) at home after passing the evaluation by a Zhan-Zhuang master
  Interventions: Other: zhan-zhuang
- Self-acupressure group (Experimental): The intervention will last 8 weeks and comprise the following
  1) Two sessions of self-acupressure training (2 hours per session/week, totally 4 hours) for 2 weeks. (2) self-practice of acupressure for 6 weeks (daily, around 20 mins) at home after passing the evaluation by a licensed traditional Chinese medicine doctor.
  Interventions: Other: self-acupressure
- Waitlist control group (No Intervention): Usual care only

INTERVENTIONS:
Other: zhan-zhuang — zhan-zhuang as a fundamental type of qigong
  Arms: Zhan-zhuang group
Other: self-acupressure — Self-acupressure as a common type of traditional Chinese medicine therapies
  Arms: Self-acupressure group

SUMMARY:
The proposed study will be a 3-arm, parallel-group randomized controlled trial on the effects of self-acupressure and Zhan-Zhuang for alleviating pain, fatigue, and sleep disturbance in breast cancer survivors. Subjects will include 54 breast cancer survivors who have experienced a moderate level of pain, fatigue and sleep disturbance. All eligible subjects will be randomized into one of the three groups in a 1:1:1 ratio: Zhan Zhuang group, or self-acupressure group, or wait list control group. Subjects in the Zhan-Zhuang group will receive up to 8 weeks of the intervention consisting of a training course over two weeks followed by self-practice for 6 weeks. Those in the self-acupressure group will attend an acupressure training course for two weeks and then, will be asked to practice self-acupressure for 6 weeks. The wait list control group will be provided with delayed self-acupressure or Zhan Zhuang at the end of the study. Outcome assessment will be conducted at baseline, week 8 (post-intervention) and week 12 (4 week follow-up). Primary outcomes include pain, fatigue and sleep disturbance. Secondary outcomes include psychological distress and health-related quality of life. Qualitative data will be collected from selected participants who have received the intervention.

ELIGIBILITY:
Inclusion Criteria:

* a female adult aged 18 and older;
* a diagnosis of early-stage (Stage I, II, or III) breast cancer;
* completion of surgery, and/or chemotherapy and/or radiotherapy;
* have at least a moderate level of pain, fatigue and sleep disturbance as measured on 0-10 numerical rating scales, with a score of ≥ 3 for each symptom during the past one month;
* willing to use WhatsApp messenger for follow-ups;
* being able to communicate in Chinese

Exclusion Criteria:

* prior use of acupuncture, acupressure, Zhan Zhuang, or other types of Zhan Zhuang within the past three months;
* currently receiving progressive muscle relaxation, mindfulness-based stress reduction, and other body mind exercise (e.g. yoga) for the treatment of pain, fatigue, and sleep disturbance;
* mentally incapable of participating in the study as indicated by the Hong Kong version of Montreal Cognitive Assessment score;
* inability to perform self-care as indicated by the Karnofsky Performance Scale score<70

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
Pain(severity and interference) | Baseline, after 8 weeks, after 12 weeks
  Pain will be measured by the traditional Chinese version of the Brief Pain Inventory. The questionnaire has 9 items assessing pain severity and interference with activities. It is rated using a 0-10 scale (0= no pain and no interference, 10=pain as bad as one can imagine and interferes completely).
Fatigue | Baseline, after 8 weeks, after 12 weeks
  Fatigue will be measured by the traditional Chinese version of the Brief Fatigue Inventory. The questionnaire has 9 items assessing pain severity and interference with activities. It is rated using a 0-10 scale (0= no pain and no interference, 10=pain as bad as one can imagine and interferes completely).
Sleep disturbance | Baseline, after 8 weeks, after 12 weeks
  Sleep disturbance will be measured by the 19-item traditional Chinese version of the Pittsburgh Sleep Quality Index. The questionnaire consists of seven domains using 19 items: overall sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, day dysfunction due to sleepiness, and use of sleeping medication. The global score is calculated by summing up the scores of seven domains, with a higher score indicating greater sleep disturbance.

SECONDARY OUTCOMES:
Psychological distress | Baseline, after 8 weeks, after 12 weeks
  Psychological distress will be measured by the 4-item traditional Chinese version of the Patient Health Questionnaire-4. The questionnaire has two subscales, with the 2-item General Anxiety Disorder screener for assessing anxiety and the 2-item Patient Health Questionnaire for assessing depression. Each item is rated on a 4-point scale ranging from 0 (not at all) to 3 (nearly every day) and the subscale scale ranges from 0 to 6.
Health-related quality of life | Baseline, after 8 weeks, after 12 weeks
  Health-related quality of life will be measured by the 27-item Traditional Chinese version of the Functional Assessment of Cancer Therapy scale. The questionnaire is a 27-item cancer-specific measure and consists of four domains: physical, social/family, emotional, and functional. Scores of items in specific domains will be created to produce subscale scores and subsequently added to produce a total scale. A higher score reflects better health-related quality of life

OTHER OUTCOMES:
Feasibility of the study | After 12 weeks
  Eligibility rate
Feasibility of the study | After 12 weeks
  Recruitment rate
Feasibility of the study | After 12 weeks
  Retention rate
Feasibility of the study | After 12 weeks
  Reasons for withdrawal from the study as collected from participants through calling them
Acceptability of the study | After 8 weeks of the intervention
  Measured by the 10-item adapted Theoretical Framework of Acceptability Questionnaire (1=disagree, 5=agree). A higher score indicates higher acceptability
Acceptability of the study | After 8 weeks of the intervention
  Qualitative in-depth interviews

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University (posters, Facebook, WhatsApp groups etc.), Hong Kong, China

IPD SHARING:
Plan to Share IPD: No